CLINICAL TRIAL: NCT01071252
Title: A Randomized, Double-blind, Placebo Controlled, Multicenter Dose Ranging Study of Subcutaneously Administered AIN457, Assessing Psoriasis Area and Severity Index (PASI) Response in Patients With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: A Dose Ranging Study of AIN457 in Patients With Moderate to Severe Chronic Plaque-type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457A2220; 2009-016807-42
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Plaque-type Psoriasis
Keywords: Moderate to severe chronic plaque-type psoriasis; AIN457; dermatology
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- AIN457 1x25mg (Experimental)
  Interventions: Drug: AIN457
- AIN457 3x25mg (Experimental)
  Interventions: Drug: AIN457
- AIN457 3x75mg (Experimental)
  Interventions: Drug: AIN457
- AIN457 3x150mg (Experimental)
  Interventions: Drug: AIN457
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIN457
  Arms: AIN457 1x25mg; AIN457 3x150mg; AIN457 3x25mg; AIN457 3x75mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether, in patients with moderate to severe plaque-type psoriasis, AIN457 administered subcutaneously reduces the severity of psoriasis symptoms and the extent to which the patient's body area is affected by the disease (compared to placebo).

ELIGIBILITY:
Inclusion Criteria:

Chronic plaque-type psoriasis diagnosed for at least 6 months at time of randomization

At randomization, moderate to severe psoriasis as defined by:

* PASI score of 12 or greater and,
* IGA score of 3 or greater and,
* Body Surface Area (BSA) affected by plaque-type psoriasis of 10% or greater At screening and randomization, chronic plaque-type psoriasis considered inadequately controlled by topical treatment.

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type
* Drug-induced psoriasis (e.g., new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium) at randomization
* Previous exposure to AIN457
* Ongoing use of prohibited psoriasis treatments / medications and other prohibited medication at randomization. Washout periods detailed in the protocol have to be adhered to
* Known immunosuppression (e.g., AIDS) at screening and / or randomization
* History or evidence of active tuberculosis at screening
* Active systemic infections (other than common cold)
* History or symptoms of malignancy of any organ system, treated or untreated, within the past 5 years.
* Any severe, progressive or uncontrolled medical condition at randomization that in the judgment of the investigator prevents the patient from participating in the study
* Any clinically significant abnormal laboratory tests at randomization, that in the judgment of the investigator prevents the patient from participating in the study
* Inability or unwillingness to undergo repeated venipuntures
* History or evidence of drug or alcohol abuse
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- United States (5):
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Lake Oswego, Oregon
  - Novartis Investigative Site, Portland, Oregon
- Canada (3):
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, North Bay, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
- Estonia (3):
  - Novartis Investigative Site, Tallinn, Estonia
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Novartis Investigative Site, Kopavogur, Iceland
- Japan (4):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Saitama, Saitama
- Novartis Investigative Site, Riga, Latvia

REFERENCES:
- See also: Click here for more information about this study: — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- AIN457 1x25mg: AIN457 25mg Subcutaneously as a single dose
- AIN457 3x25mg: AIN457 25mg subcutaneous monthly dosing, 3 times (weeks 1, 5, and 9)
- AIN457 3x75mg: AIN457 75mg subcutaneous monthly dosing, 3 times (weeks 1, 5, and 9)
- AIN457 3x150mg: AIN457 150mg subcutaneous monthly dosing, 3 times (weeks 1, 5, and 9)
- Placebo: Placebo subcutaneous monthly dosing, 3 times (weeks 1, 5, and 9)
Period: Overall Study
Arm/Group | AIN457 1x25mg | AIN457 3x25mg | AIN457 3x75mg | AIN457 3x150mg | Placebo
Started | 29 | 26 | 21 | 27 | 22
Completed | 14 | 16 | 17 | 20 | 11
Not Completed | 15 | 10 | 4 | 7 | 11
Not completed — unsatisfactory therapeutic effect | 4 | 6 | 2 | 0 | 6
Not completed — Withdrawal by Subject | 8 | 2 | 1 | 2 | 3
Not completed — administrative problems | 1 | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 1x25mg | AIN457 3x25mg | AIN457 3x75mg | AIN457 3x150mg | Placebo | Total
Number analyzed (Participants) | 29 | 26 | 21 | 27 | 22 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (12.65) | 46.3 (13.43) | 45.8 (12.36) | 45.4 (11.64) | 45.9 (10.88) | 45.9 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 7 | 6 | 8 | 34
  Male | 20 | 22 | 14 | 21 | 14 | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants of Reponders of Psoriasis Area and Severity Index (PASI) 75 Achievement at Week 13
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: week 13
Population: The full analysis set (FAS), identical to the randomized set, also consisted of all randomized patients.
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 1x25mg | AIN457 3x25mg | AIN457 3x75mg | AIN457 3x150mg | Placebo
Number analyzed (Participants) | 29 | 26 | 21 | 27 | 22
percentage of participants | 3.4 | 19.2 | 57.1 | 81.5 | 9.1

2. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Response
Description: IGA treatment response is defined as achievement of IGA 0 (clear) or 1 (almost clear) and improvement of at least 2 points on the IGA scale compare with baseline.
Time Frame: Week 2, 3, 5, 9, 13, 17, 21, 25, 29, 33, 37
Population: The full analysis set (FAS), identical to the randomized set, also consisted of all randomized patients.
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 1x25mg | AIN457 3x25mg | AIN457 3x75mg | AIN457 3x150mg | Placebo
Number analyzed (Participants) | 29 | 26 | 21 | 27 | 22
percentage of participants
  Week 2 | 0 | 0 | 0 | 3.7 | 0
  Week 3 | 0 | 0 | 0 | 3.7 | 0
  Week 5 | 0 | 3.8 | 4.8 | 7.4 | 0
  Week 9 | 0 | 7.7 | 28.6 | 37 | 9.1
  Week 13 | 0 | 11.5 | 33.3 | 48.1 | 9.1
  Week 17 | 3.4 | 19.2 | 28.6 | 51.9 | 9.1
  Week 21 | 0 | 19.2 | 38.1 | 40.7 | 13.6
  Week 25 | 0 | 15.4 | 33.3 | 37 | 18.2
  Week 29 | 0 | 11.5 | 19.0 | 40.7 | 13.6
  Week 33 | 0 | 15.4 | 19.0 | 29.6 | 0
  Week 37 | 0 | 15.4 | 9.5 | 25.9 | 0

3. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI 50, PASI 75 or PASI 90)
Description: as for outcome 1
Time Frame: Week 2, 3, 5, 9, 13, 17, 21, 25, 29, 33, 37
Population: The full analysis set (FAS), identical to the randomized set, also consisted of all randomized patients.
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN457 1x25mg | AIN457 3x25mg | AIN457 3x75mg | AIN457 3x150mg | Placebo
Number analyzed (Participants) | 29 | 26 | 21 | 27 | 22
Percentage of Participants
  Week 2 PASI 50 | 3.4 | 7.7 | 4.8 | 11.1 | 0
  Week 2 PASI 75 | 0 | 0 | 0 | 0 | 0
  Week 2 PASI 90 | 0 | 0 | 0 | 0 | 0
  Week 3 PASI 50 | 3.4 | 7.7 | 23.8 | 18.5 | 4.5
  Week 3 PASI 75 | 0 | 0 | 0 | 0 | 0
  Week 3 PASI 90 | 0 | 0 | 0 | 0 | 0
  Week 5 PASI 50 | 10.3 | 15.4 | 28.6 | 48.1 | 4.5
  Week 5 PASI 75 | 0 | 7.7 | 4.8 | 14.8 | 4.5
  Week 5 PASI 90 | 0 | 0 | 0 | 3.7 | 0
  Week 9 PASI 50 | 10.3 | 38.5 | 52.4 | 85.2 | 13.6
  Week 9 PASI 75 | 3.4 | 11.5 | 33.3 | 66.7 | 9.1
  Week 9 PASI 90 | 0 | 3.8 | 9.5 | 14.8 | 0
  Week 13 PASI 50 | 17.2 | 57.7 | 81.0 | 85.2 | 18.2
  Week 13 PASI 75 | 3.4 | 19.2 | 57.1 | 81.5 | 9.1
  Week 13 PASI 90 | 0 | 7.7 | 19.0 | 51.9 | 4.5
  Week 17 PASI 50 | 20.7 | 53.8 | 76.2 | 85.2 | 27.3
  Week 17 PASI 75 | 6.9 | 26.9 | 42.9 | 81.5 | 13.6
  Week 17 PASI 90 | 0 | 15.4 | 9.5 | 44.4 | 0
  Week 21 PASI 50 | 13.8 | 50.0 | 57.1 | 85.2 | 31.8
  Week 21 PASI 75 | 0 | 23.1 | 38.1 | 77.8 | 13.6
  Week 21 PASI 90 | 0 | 15.4 | 9.5 | 37.0 | 4.5
  Week 25 PASI 50 | 13.8 | 50.0 | 57.1 | 85.2 | 31.8
  Week 25 PASI 75 | 0 | 19.2 | 33.3 | 70.4 | 9.1
  Week 25 PASI 90 | 0 | 11.5 | 19.0 | 29.6 | 4.5
  Week 29 PASI 50 | 17.2 | 46.2 | 52.4 | 85.2 | 27.3
  Week 29 PASI 75 | 0 | 15.4 | 23.8 | 59.3 | 13.6
  Week 29 PASI 90 | 0 | 7.7 | 14.3 | 22.2 | 9.1
  Week 33 PASI 50 | 10.3 | 34.6 | 47.6 | 77.8 | 22.7
  Week 33 PASI 75 | 3.4 | 19.2 | 23.8 | 55.6 | 4.5
  Week 33 PASI 90 | 0 | 0 | 9.5 | 18.5 | 4.5
  Week 37 PASI 50 | 17.2 | 30.8 | 47.6 | 63.0 | 22.7
  Week 37 PASI 75 | 3.4 | 19.2 | 19.0 | 25.9 | 4.5
  Week 37 PASI 90 | 0 | 3.8 | 9.5 | 11.1 | 4.5

4. Secondary Outcome: To Assess the Time to Relapse
Description: Relapse is defined as the loss of at least 50% of the maximum PASI change from baseline achieved at any time before that visit and analyzed only for the active treatment groups.
Time Frame: 37 weeks
Population: The full analysis set (FAS), identical to the randomized set, also consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AIN457 1x25mg | AIN457 3x25mg | AIN457 3x75mg | AIN457 3x150mg
Number analyzed (Participants) | 1 | 5 | 12 | 22
days | NA [NA to NA] — Not Estimable because no relapses occured | NA [NA to NA] — Not Estimable because no relapses occured | NA [198 to NA] — Not Estimable because very low relapses occured | 203 [203 to NA] — Not Estimable because very low relapses occured

ADVERSE EVENTS:
Arm/Group | AIN457 1x25mg | AIN457 3x25mg | AIN457 3x75mg | AIN457 3x150mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/29 | 2/26 | 1/21 | 0/27 | 2/22
Other Adverse Events (participants affected / at risk) | 14/29 | 11/26 | 10/21 | 16/27 | 8/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 1x25mg (N=29) | AIN457 3x25mg (N=26) | AIN457 3x75mg (N=21) | AIN457 3x150mg (N=27) | Placebo (N=22)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 1x25mg (N=29) | AIN457 3x25mg (N=26) | AIN457 3x75mg (N=21) | AIN457 3x150mg (N=27) | Placebo (N=22)
Fatigue (General disorders) | 0 | 0 | 0 | 3 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 4 | 4 | 4 | 2
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 1 | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 1 | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 8 | 4 | 4 | 3 | 2
Hypertension (Vascular disorders) | 1 | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.